CLINICAL TRIAL: NCT05233098
Title: TheraSphere Post-approval Study to Calculate the Radiation-absorbed Dose of Technetium-99m Macroaggregated Albumin (Tc-99m MAA) to the Whole Body and Non-liver Critical Organs.
Brief Title: TheraSphere Post-Approval Study to Calculate the Radiation-absorbed Dose of Tc-99m MAA.
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2494
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma; Carcinoma, Hepatocellular; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Clinical Cohort: Patients enrolled in the study will have 3 imaging scans taken after Tc-99m MAA injection. The final scan will occur between 18 and 24 hours after Tc-99m MAA injection.
  Interventions: Device: Technetium-99m macroaggregated albumin (Tc-99m MAA)

INTERVENTIONS:
Device: Technetium-99m macroaggregated albumin (Tc-99m MAA) — Patients who are being evaluated for TheraSphere administration.

SUMMARY:
The TheraSphere Post-Approval Study is a post-market, prospective, single-arm, open-label, observational study to support the use of TheraSphere for the treatment of hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Every patient being treated with TheraSphere needs to have a screening procedure with the administration of a radioactive product named Tc-99m MAA (called pre-treatment mapping). This screening procedure aims to determine if the patient can be treated with TheraSphere. The purpose of this study is to better understand the dose of radiation that is absorbed by the body and the risk of Tc-99m MAA to the whole body and other organs around the liver. The study will determine the amount of Tc-99m MAA that stays in the body and organs up to 24 hours after the administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21 years and older
2. Written informed consent
3. Patients who receive Tc-99m MAA while being evaluated for TheraSphere treatment.

Exclusion Criteria:

1. Patients who are contraindicated for TheraSphere treatment.
2. Patients who are contraindicated for Tc-99m MAA per the applicable Package Insert.
3. Patients who do not receive Tc-99m MAA during pre-treatment Y-90 mapping

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The intended population for the TheraSphere Post-Approval study is patients with HCC who are undergoing evaluation to assess eligibility for TheraSphere treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical study site, NWU in Chicago, IL USA. Six patients consented and enrolled. Patient considered enrolled at time of consent per protocol. Patient 001 withdrew consent prior to the Tc-99m MAA procedure. Five patients received protocol required imaging after Tc-99m MAA injections.
  Patient # Date of Enrollment:
  1. Apr 4, 2022
  2. Feb 4, 2023
  3. Mar 4, 2023
  4. Mar 14, 2023
  5. May 10, 2023
  6. Jun 6, 2023
Period: Overall Study
Arm/Group | Clinical Cohort
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Participants.: Female | 1
  Participants.: Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Whole Body
Description: To provide imaging data calculating radiation-delivered dose of Tc-99m MAA to the whole body.
Time Frame: Immediately following
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Groups:
- Clinical Cohort: First imaging scan taken after Tc-99m MAA injection.
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 67.322 [43.22 to 85.50]

2. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Non-Liver Critical Organs
Description: To provide imaging data to calculate the radiation-delivered dose of Tc-99m MAA to the whole body and to potential irradiated non-liver critical organs.
Time Frame: Immediately following
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 6.986 [2.91 to 12.32]

3. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Whole Body
Description: To provide imaging data to calculate the radiation-delivered dose of Tc-99m MAA to the whole body.
Time Frame: 4 hours +/- 2 hours
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 27.978 [16.22 to 36.20]

4. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Non-Liver Critical Organs.
Description: as for outcome 2
Time Frame: 4 hours +/- 2 hours
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 8.640 [4.57 to 14.01]

5. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Whole Body.
Description: To provide imaging data calculating radiation-delivered dose of Tc-99m MAA to the whole body following injection.
Time Frame: 18-24 hours
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 1.694 [0.25 to 3.90]

6. Primary Outcome: Delivered Activity of Tc-99m MAA (MBq) for Non-Liver Critical Organs
Description: To provide imaging data to calculate radiation delivered dose of Tc-99m MAA to the whole body and to potential irradiated non-liver critical organs.
Time Frame: 18-24 hours
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: MBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
MBq | 0.662 [0.11 to 1.64]

7. Primary Outcome: Absorbed Dose of Tc-99m MAA (mGy) for Whole Body.
Description: To provide imaging data calculating radiation-absorbed dose of Tc-99m MAA to the whole body.
Time Frame: Overall
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: mGy
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
mGy | 10.970 [9.950 to 11.310]

8. Primary Outcome: Absorbed Dose of Tc-99m MAA (mGy) for Non-Liver Critical Organs
Description: To provide imaging data calculating radiation-absorbed dose of Tc-99m MAA to Non-Liver Critical Organs.
Time Frame: Overall
Population: Patient who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: mGy
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
mGy | 4.812 [2.68 to 8.05]

9. Primary Outcome: Effective Dose of Tc-99m MAA (mSv) Whole Body
Description: To provide imaging data calculating radiation-effective does of Tc-99m MAA to Non-Liver Critical Organs.
Time Frame: Overall
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: mSv
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
mSv | 0.666 [0.56 to 0.78]

10. Primary Outcome: Effective Dose of Tc-99m MAA (mSv/mBq) for Whole Body
Description: To provide data calculating radiation-effective dose of Tc-99m MAA to Whole Body.
Time Frame: Overall
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Median (Inter-Quartile Range); unit: mSv/mBq
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
mSv/mBq | 0.008 [0.008 to 0.008]

11. Primary Outcome: Equivalent Dose of TC-99m MAA (mSV) for Non-Liver Critical Organs
Description: To provide imaging data calculating radiation-equivalent dose of Tc-99m MAA to Non-Liver Critical Organs.
Time Frame: Overall
Population: Patients who are being evaluated for TheraSphere administration.
Measure: Mean (Full Range); unit: mSv
Arm/Group | Clinical Cohort
Number analyzed (Participants) | 5
mSv | 0.384 [0.10 to 0.65]

ADVERSE EVENTS:
Time Frame: Procedure-related Serious Adverse Events were assessed immediately following Tc-99m MAA injection, 4 hours (+ or = to 2 hours) following Tc-99m MAA injection, > or = to 18 hours but < or = to 24 hours following Tc-99m MAA injection.
Arm/Group | Clinical Cohort
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT05233098/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT05233098/SAP_001.pdf